CLINICAL TRIAL: NCT05697419
Title: Integrating NIH Reset Stress Strategies Into DPT Curriculum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Shannon Dudash, Doctor of Physical Therapy, Youngstown State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-155
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Stress
MeSH Terms: interventions — Muscle Relaxation; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DPT students at YSU (Other)
  Interventions: Behavioral: deep breathing, muscle relaxation, and mindfulness

INTERVENTIONS:
Behavioral: deep breathing, muscle relaxation, and mindfulness — 5-10-minute group sessions will be administered to DPT students teaching them the NIH recommended strategies of deep breathing, muscle relaxation or mindfulness.

SUMMARY:
The goal of this longitudinal prospective cohort study is to determine effectiveness of integrating NIH reset stress strategies of deep breathing, muscle relaxation and mindfulness in DPT students in order to help them reduce stress throughout their schooling.

The main question[s] it aims to answer are:

* Do performing the NIH reset stress strategies help DPT students manage their stress
* Do DPT students find these strategies helpful Participants will be asked to fill out initial intake forms and participate in weekly sessions of five to ten minutes that will be either a deep breathing, mindfulness, or muscle relaxation activity led by faculty member. DPT students will then rate their stress level weekly on a numeric stress scale.

DETAILED DESCRIPTION:
Integrating NIH Reset Stress Strategies into DPT Curriculum A. Investigator Information

1. Primary Investigator: Shannon Dudash PT, DPT, GCS
2. Co-Investigators: Weiqing Ge PhD, PT, Nancy Landgraff PhD, PT, Cara Berg-Carramusa EdD, PT B. Sponsor/Funding Information

a. Not applicable C. Location of Research

a. Youngstown State University D. Conflict of Interest

a. none E. Methods and Procedures

a. Introduction i. DPT students report higher levels of stress and anxiety compared to their age matched peers (1). Since 2020, COVID has caused increased stress among students and the general population (11, 12). Increased stress can negatively impact not only students' physical conditions but also their academic performance. This may potentially have long term consequences that carry over into their careers and lead to decreased quality of future healthcare workers. There is a lack of information on if and how DPT programs address stress in DPT students in their curriculum. Deep breathing, muscle relaxation and mindfulness are strategies recommended by the NIH to help manage stress to general public which can potentially be used by DPT program to help DPT students manage their stress and be successful. However, there is lack of evidence on the use of these strategies to assist DPT students manage stress and anxiety during their schooling.

b. Background i. Long term stress, or chronic stress, can lead to serious health problems including disrupted sleep, muscle tension, metabolic dysfunction, immune abnormalities, and inflammation. Some diseases such as cardiovascular disease, diabetes, cancer, autoimmune diseases, depression, and anxiety orders can be linked to chronic stress.

ii. Deep breathing, mindfulness, and muscle relaxation have been used to manage stress in older and younger adult populations (3, 4, 6, 13).

c. Objectives i. The purpose of this study is to determine the effectiveness of integrating NIH reset stress strategies of deep breathing, muscle relaxation and mindfulness for DPT students in order to help them reduce stress throughout their schooling.

d. Study design and procedures i. How the participants will be identified and recruited and how informed consent will be obtained to minimize coercion or undue influence: The study design is a longitudinal prospective cohort study. Students in the Doctor of Physical Therapy program will be recruited by email about the "Integrating NIH Reset Stress Strategies into DPT Curriculum" project, NIH Reset Stress flyer, and an informed consent form from the student worker in the Graduate of Health Sciences department. A recruitment flyer will be posted within the department. Also, a current student will recruit within the DPT classes. If students choose to participate, they will turn in their signed informed consent to Shannon Dudash by the end of week 1 of the spring semester.

ii. Procedures for data collection: Initial meeting will be established with participants to fill out intake paperwork including survey asking if participants know what deep breathing, muscle relaxation, and mindfulness are, demographic information, DASS-21, PSS-10 and Stress Numeric Scale.

iii. Procedures to which human subjects will be exposed: Reset Stress sessions will be administered prior to the start of a weekly class by the course instructor (Shannon Dudash). The focus of the sessions will be a combination of mindfulness, deep breathing, and muscle relaxation. These sessions will last approximately 5-10 minutes. Sessions will be performed in a group setting. There will be a total of 12-14 sessions administered throughout the 2023 Spring semester at YSU on a weekly basis.

iv. Procedures for data collection: Participants will fill out a Stress Numeric Scale after each weekly intervention session. Participants will also be asked to complete the DASS-21, Stress Numeric Scale, and PSS-10 at a midpoint check-in during week 6 and at the end of the project. An additional survey at the end of the project inquiring if it was helpful to learn these stress management strategies and how frequently participants used them independently will be administered.

v. Any paper forms used will not have any identification on them to protect participant privacy. Anonymous Slido presentation will be used to collect weekly Stress Numeric scale ratings.

vi. Data Analysis will include comparison of surveys from start to completion of sessions. We will use a repeated measure ANOVA to look at trends of Stress Numeric scale over the spring semester. Descriptive analysis will also include participants' responses on how frequently they used the stress management strategies independently and if they found that the strategies taught were beneficial.

e. No deception is to be used in this study. f. Participants will not be presented with materials that they might regard to be offensive, threatening or degrading.

F. Risk/Benefit Assessment a. Potential risks: It is unlikely, but the participants might have negative feelings by recalling previous experience when completing the questionaries. It will be no more than what they feel in normal daily life.

G. Potential benefits: Benefits from this study include learning different strategies to control stress. Implementing the strategies may reduce stress, improve physical conditions, and improve academic performance.

H. Human Research Participants

a. Students enrolled in Doctor of Physical Therapy program at Youngstown State University i. Inclusion criteria: age > 18 years old, enrolled in DPT program ay YSU, ability to follow instructions to perform deep breathing, muscle relaxation, and mindfulness strategies.

ii. Exclusion criteria: age < 18 years old, not enrolled in DPT program at YSU I. Recruitment Procedures

1. Students in the Doctor of Physical Therapy program will be recruited by email about the "Integrating NIH Reset Stress Strategies into DPT Curriculum" project, NIH Reset Stress flyer and an informed consent form from the student worker in the Graduate of Health Sciences department. A recruitment flyer will be posted within the department. Also, a current student will recruit within the DPT classes.
2. If students choose to participate, they will turn in their signed informed consent to Shannon Dudash by the end of week 1 of the spring semester.

J. Informed Consent and Assent

1. Informed consent attached to IRB application separately
2. No minors, prisoners, or individuals with intellectual disabilities will be included in this study.
3. The record of informed consent will be stored in the principal investigator's office in a locked filing cabinet.

K. Confidentiality of Information Collected

1. All outcome measures will be collected anonymously. No names of the participants will be collected except the informed consent form.
2. Data will be stored on Research laptop computer that is password protected. All signed informed consent forms will be stored in a locked file cabinet in a locked office on Youngstown State University Campus and will be shredded after 3 years in accordance with IRB standards.

ELIGIBILITY:
Inclusion Criteria:

* DPT student at Youngstown State University
* > 18 years old
* Have the ability to follow instructions to perform deep breathing, muscle relaxation, and mindfulness strategies

Exclusion Criteria:

* Not a DPT student at Youngstown State University
* Under 18 years of age

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
PSS-10 | through study completion, an average of 1 year
  Stress questionnaire
DASS-21 | through study completion, an average of 1 year
  Depression, stress and Anxiety questionnaire

SECONDARY OUTCOMES:
Stress Numeric scale | through study completion, an average of 1 year
  1 through 10 scale rating stress level from nothing to extremely high

CONTACTS AND LOCATIONS:
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gallego-Gomez JI, Balanza S, Leal-Llopis J, Garcia-Mendez JA, Oliva-Perez J, Domenech-Tortosa J, Gomez-Gallego M, Simonelli-Munoz AJ, Rivera-Caravaca JM. Effectiveness of music therapy and progressive muscle relaxation in reducing stress before exams and improving academic performance in Nursing students: A randomized trial. Nurse Educ Today. 2020 Jan;84:104217. doi: 10.1016/j.nedt.2019.104217. Epub 2019 Oct 18. PMID 31683132
- [Result] Lesage FX, Berjot S, Deschamps F. Clinical stress assessment using a visual analogue scale. Occup Med (Lond). 2012 Dec;62(8):600-5. doi: 10.1093/occmed/kqs140. Epub 2012 Sep 10. PMID 22965867
- [Result] Perciavalle V, Blandini M, Fecarotta P, Buscemi A, Di Corrado D, Bertolo L, Fichera F, Coco M. The role of deep breathing on stress. Neurol Sci. 2017 Mar;38(3):451-458. doi: 10.1007/s10072-016-2790-8. Epub 2016 Dec 19. PMID 27995346
- [Result] Gardi C, Fazia T, Stringa B, Giommi F. A short Mindfulness retreat can improve biological markers of stress and inflammation. Psychoneuroendocrinology. 2022 Jan;135:105579. doi: 10.1016/j.psyneuen.2021.105579. Epub 2021 Nov 6. PMID 34775250
- [Result] Pascoe MC, Thompson DR, Jenkins ZM, Ski CF. Mindfulness mediates the physiological markers of stress: Systematic review and meta-analysis. J Psychiatr Res. 2017 Dec;95:156-178. doi: 10.1016/j.jpsychires.2017.08.004. Epub 2017 Aug 23. PMID 28863392
- [Result] Pascoe MC, Thompson DR, Ski CF. Yoga, mindfulness-based stress reduction and stress-related physiological measures: A meta-analysis. Psychoneuroendocrinology. 2017 Dec;86:152-168. doi: 10.1016/j.psyneuen.2017.08.008. Epub 2017 Aug 30. PMID 28963884
- [Result] Zhang L, Qi H, Wang L, Wang F, Huang J, Li F, Zhang Z. Effects of the COVID-19 pandemic on acute stress disorder and career planning among healthcare students. Int J Ment Health Nurs. 2021 Aug;30(4):907-916. doi: 10.1111/inm.12839. Epub 2021 May 17. PMID 34002465
- [Result] Wang C, Wen W, Zhang H, Ni J, Jiang J, Cheng Y, Zhou M, Ye L, Feng Z, Ge Z, Luo H, Wang M, Zhang X, Liu W. Anxiety, depression, and stress prevalence among college students during the COVID-19 pandemic: A systematic review and meta-analysis. J Am Coll Health. 2023 Oct;71(7):2123-2130. doi: 10.1080/07448481.2021.1960849. Epub 2021 Sep 1. PMID 34469261
- [Result] Heckenberg RA, Eddy P, Kent S, Wright BJ. Do workplace-based mindfulness meditation programs improve physiological indices of stress? A systematic review and meta-analysis. J Psychosom Res. 2018 Nov;114:62-71. doi: 10.1016/j.jpsychores.2018.09.010. Epub 2018 Sep 22. PMID 30314581
- See also: Depression, stress and anxiety in DPT students — https://doi.org/10.1097/jte.0000000000000185
- See also: Perfectionism, Stress, and the Entry-Level Doctor of Physical Therapy Student — https://doi.org/10.1097/JTE.0000000000000213